CLINICAL TRIAL: NCT00599846
Title: The Natural History of Geographic Atrophy Progression (GAP) Study
Status: Terminated | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Patricia Zilliox, Alcon
Other Study IDs: C-06-30
Record Dates: First submitted 2008-01-13; First posted 2008-01-24 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Age-Related Macular Degeneration; Geographic Atrophy
Keywords: age-related macular degeneration; geographic atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the 18-month trial is to evaluate the natural history of geographic atrophy by assessing the rate of progression of the geographic atrophic lesion over time.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of geographic atrophy secondary to age-related macular degeneration with no CNV lesion.

Exclusion Criteria:

* Age related

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients showing signs of geographic atrophy secondary to age-related macular degeneration with no CNV lesion.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
GA progression rate using fundus autofluorescence | From baseline

SECONDARY OUTCOMES:
GA progression rate using fundus photography | From baseline

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Zilliox, Study Director — Alcon Research
Locations (1):
- Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Steinberg JS, Auge J, Jaffe GJ, Fleckenstein M, Holz FG, Schmitz-Valckenberg S; GAP Study Group. Longitudinal analysis of reticular drusen associated with geographic atrophy in age-related macular degeneration. Invest Ophthalmol Vis Sci. 2013 Jun 10;54(6):4054-60. doi: 10.1167/iovs.12-11538. PMID 23633663
- [Derived] Mauschitz MM, Fonseca S, Chang P, Gobel AP, Fleckenstein M, Jaffe GJ, Holz FG, Schmitz-Valckenberg S; GAP Study Group. Topography of geographic atrophy in age-related macular degeneration. Invest Ophthalmol Vis Sci. 2012 Jul 26;53(8):4932-9. doi: 10.1167/iovs.12-9711. PMID 22661483
- [Derived] Schmitz-Valckenberg S, Alten F, Steinberg JS, Jaffe GJ, Fleckenstein M, Mukesh BN, Hohman TC, Holz FG; Geographic Atrophy Progression (GAP) Study Group. Reticular drusen associated with geographic atrophy in age-related macular degeneration. Invest Ophthalmol Vis Sci. 2011 Aug 24;52(9):5009-15. doi: 10.1167/iovs.11-7235. PMID 21498612
- [Derived] Schmitz-Valckenberg S, Fleckenstein M, Gobel AP, Hohman TC, Holz FG. Optical coherence tomography and autofluorescence findings in areas with geographic atrophy due to age-related macular degeneration. Invest Ophthalmol Vis Sci. 2011 Jan 5;52(1):1-6. doi: 10.1167/iovs.10-5619. PMID 20688734